CLINICAL TRIAL: NCT07271641
Title: Clinical and Microbial Evaluation of Two Different Implant Retained Mandibular Overdentures (Randomized Clinical Trial)
Brief Title: A Study Comparing Two Different Denture Base Materials in Implant Retained Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Noha Taha Kamel Taha Alloush, Lecturer, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29.4.24
Record Dates: First submitted 2025-11-18; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Edentulous Alveolar Ridge In Mandible; Edentulous Jaw; Edentulous Mouth; Implant Supported Overdenture; Attachments; Dental Implant; Complete Edentulism
Keywords: Dental Implants; Completely edentulous patients; Edentulous Ridge; Candida; Patient Satisfaction; Clinical Parameters
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous; Torulopsis; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mandibular complete dentures processed into heat cured acrylic resin (Active Comparator): mandibular complete dentures made of heat-cured acrylic resin polymethylmethacrylate (PMMA). In the mandible, two implants were inserted in the symphyseal area and retained by Novaloc attachments.
  Interventions: Procedure: Conventional acrylic resin denture
- mandibular thermoplastic nylon denture (Experimental): mandibular overdentures were made of the flexible acrylic resin breflex, In the mandible, two implants were inserted in the symphyseal area and retained by Novaloc attachments.
  Interventions: Procedure: Flexible resin denture

INTERVENTIONS:
Procedure: Conventional acrylic resin denture — Mandibular complete dentures made of heat-cured acrylic resin polymethylmethacrylate (PMMA). In the mandible, two implants were inserted in the symphyseal area and retained by Novaloc attachments.
  Arms: mandibular complete dentures processed into heat cured acrylic resin
Procedure: Flexible resin denture — Mandibular overdentures were made of the flexible acrylic resin breflex, In the mandible, two implants were inserted in the symphyseal area and retained by Novaloc attachments
  Arms: mandibular thermoplastic nylon denture

SUMMARY:
The aim of removable prosthodontics is not only to restore lost oral structures but also to preserve the remaining tissues. Implant-retained overdentures have shown superior outcomes over conventional dentures by reducing residual ridge resorption, enhancing prosthesis support and retention, and improving patients' quality of life. Retention can be further optimized through the use of various attachment systems such as bars, studs, magnets, and telescopic crowns.

Traditional PMMA denture bases have limited flexibility, making their extension into soft-tissue undercuts challenging. The introduction of flexible resin materials has improved adaptation to deeper undercuts, enhancing retention while minimizing patient discomfort and absorbing functional stresses. Additionally, flexible resins may reduce microbial colonization by improving blood circulation to the underlying mucosa and supporting salivary defense mechanisms against Candida albicans.

Recently, innovative attachment systems such as Novaloc have been developed, featuring PEEK retentive caps and an amorphous diamond-like carbon coating to minimize wear and maintain long-term retention. Their versatile design allows better accommodation of gingival variations and contributes to improved patient satisfaction and treatment success.

DETAILED DESCRIPTION:
The present study will be performed to compare the difference in microbial accumulation, quality of life and patient satisfaction for implant retained mandibular overdenture using both conventional PMMA and flexible denture base materials.

16 Patients will be equally divided into two treatment groups: Group 1: Each patient in this group will receive conventional maxillary and mandibular complete dentures made of heat-cured acrylic resin. In the mandible, two implants were inserted and retained by Novaloc attachments. Group 2: Patients in this group will receive the same type of treatment as the patients in group1 but the mandibular overdentures were made of the flexible acrylic resin

ELIGIBILITY:
Inclusion Criteria:

1. Edentulous patients were chosen between the ages of 60 to 70 years old
2. All patients' ridges were covered with firm mucosa,
3. free from any signs of inflammation or ulceration, exhibit adequate height and width of the residual alveolar ridge have sufficient inter arch space.
4. Patients were free from any metabolic or bone disorder that contraindicate implant installation.

Exclusion Criteria:

1. Patients with oral or systemic diseases
2. patients with xerostomia or excessive salivation.
3. Patients with parafunctional habits (bruxism or clenching) or history of temporo-mandibular dysfunction or brain disorders or psychiatric disorders.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Pocket depth (Depth of gingival sulcus) | Follow up visits were scheduled at denture insertion, 6, and 12 months
  The depth of the gingival sulcus will be measured around each implant using a graduated periodontal probe. This probe will be inserted between the oral sulcular epithelium and the implant with minimal pressure. The distance from the tip of the probe and the free gingival margin will be measured and recorded to the nearest millimeter. Four readings were recorded at the middle of the four surfaces, buccal, lingual, mesial, and distal. The mean of the four readings will be considered as the pocket depth for this group at the chosen time.
Plaque index | Follow up visits were scheduled at denture insertion, 6, and 12 months
  Amount of plaque accumulation was graded from (0 to 3) where: Grade 0: No plaque detected by passing the side of probe along the implant. Grade 1: Film of plaque detected by probing. Grade 2: Moderate accumulation of soft debris, which can be seen by the naked eye. Grade 3: Too much soft matter within the sulcus, gingival margin, and adjacent implant surface. For each group, four readings were recorded at the middle of the four surfaces, buccal, lingual, mesial, and distal. The mean of the four readings was considered as the plaque index for this group at the chosen times

SECONDARY OUTCOMES:
isolation of Candida albicans | Follow up visits were scheduled at denture insertion, 6, and 12 months
  A sterile swab will be rubbed on the intaglio surface of the denture. The swab will be placed in a tube containing 1 ml phosphate buffered saline solution and sonicated for 5 minutes at 35 kHz. - Serial decimal dilutions (100 to 10-2)will be prepared from the sonicated swab solution. - 100 µl of the sonicated solution will be inoculated on Sabouraud's dextrose agar at 37°C for 48 hours. - After incubation, the agar plate will be retrieved, and the number of colonies will be counted and tabulated for statistical analysis
Patient satisfaction (Questionnaire) | Follow up visits were scheduled at denture insertion, 6, and 12 months.
  Participant satisfaction will be measured using a visual analog scale (VAS) questionnaire. The questions include the appearance, ease of cleaning, speaking ability, eating comfort, and overall satisfaction of their dentures.
  Participants will marked the amount of satisfaction on a 100-mm-length line (0 = no satisfaction at all and 100 = complete satisfaction). At a location that corresponded to the subject's subjective emotion, a pencil mark was drawn across the horizontal line. The distance in millimeters between the left end limit and the pencil mark point, which represents the subject's VAS score, will then be used to calculate satisfaction. The subject's perception of the prosthesis improves with a higher score. Using the VAS scores, satisfaction levels were categorized as follows: completely unsatisfied (0-31), somewhat unhappy (>31-50), slightly satisfied (>50-79), and satisfied (>79). The questionnaire was given to the patients in Arabic
Oral Health-Related Quality of Life (OHRQoL) (Questionnaire) | Follow up visits were scheduled at denture insertion, 6, and 12 months
  The oral health impact profile (OHIP-14) questions will be utilized to assess OHRQoL. The questions are composed of seven domains: functional limitations (pronouncing sounds, sense of taste), physical pains (painful aching, comfort on eating), psychologic discomforts (self-consciousness, feeling tense), physical disabilities (unsatisfactory diet, interrupting meals), psychologic disabilities (difficult to relax, embarrassment), social disabilities (irritability with people, difficulty in jobs), and handicapping (life in general, inability to function). The responses for questions are never (=1), hardly ever (=2), occasionally (=3), fairly often (=4), and very often (=5). Lower scores indicate increased satisfaction, and higher scores indicate decreased satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Clinical Study Report
Supporting Information: Study Protocol, CSR
Time Frame: Start Date: After publication End Date: 3 years
Access Criteria: After publication through the corresponding author